CLINICAL TRIAL: NCT02282943
Title: Carbon Dioxide-laser Versus Harmonic Scalpel in the Treatment of Pelvic Pain Due to Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mr Andrew Kent (Other)
Responsible Party: Sponsor-Investigator, Mr Andrew Kent, Consultant Gynaecologist, Royal Surrey County Hospital NHS Foundation Trust
Organization: Royal Surrey County Hospital NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC71/02
Record Dates: First submitted 2014-10-30; First posted 2014-11-05 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Endometriosis
Keywords: endometriosis; CO2 laser vapourisation; Harmonic scalpel; AFS stage I-III
MeSH Terms: conditions — Endometriosis | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser (Active Comparator): vapourisation/excision of endometriosis using CO2 laser
  Interventions: Device: Laser
- Harmonic scalpel (Experimental): excision of endometriosis using Harmonic scalpel
  Interventions: Device: Harmonic scalpel

INTERVENTIONS:
Device: Laser — Vapourisation/excision of endometriosis AFS stages I-III using CO2 laser
  Arms: Laser
Device: Harmonic scalpel — Excision of endometriosis using Harmonic scalpel
  Arms: Harmonic scalpel

SUMMARY:
The purpose of this study is to compare laser CO2 ablation/excision of Endometriosis (AFS stages 1-3) with excision of endometriosis using the Ethicon Harmonic ACE device. Pain scores at 6 months was the primary outcome, but secondary outcomes assessed pain scores at 1, 3 and 5 years as well as psychological state and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis grade I-III by revised American Fertility Society Scoring
* Patients in whom laser treatment to the endometriosis is considered the treatment of choice.
* Patients having consented to participated in the trial
* Patient is 18 years old or greater
* Patients who have no contraindications to either of the treatment modalities proposed

Exclusion Criteria:

* Patients who do not wish to participate/have not signed the informed consent form
* Pregnancy of breast feeding
* Patients who are unable or unwilling to discontinue hormonal treatment for 6 months
* Patients who have received additional treatment for their endometriosis within 6 months of surgery
* Patients with documented painful conditions of the gastrointestinal or urinary system

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2002-10; Primary Completion 2011-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain score (VAS) change at 6 months compared to preoperative baseline | 6 months

SECONDARY OUTCOMES:
Quality of life survey (Endometriosis Health Profile Questionnaire) | 0, 3, 6 months and 1,3,5 years
Psychological state | 0, 3 ,6 months and 1,3,5 years
  Hospital Anxiety & Depression Scale
Visual analogue pain score (VAS) change from baseline | 1,3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kent, MD FRCOG, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust